CLINICAL TRIAL: NCT05270382
Title: Clinical Research Study to Evaluate the Effect of Colgate Mouthwashes on Oral Microbiome in Oral Tissue Samples
Brief Title: Effect of Mouthwashes on Oral Wound Healing and Microbiome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Praveen Kumar Gajendrareddy, Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2018-1417; CRO-2018-SAL-08-MW-DC (Other: Colgate-Palmolive Company)
Record Dates: First submitted 2021-12-07; First posted 2022-03-08 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Wound Heal; Oral Microbiome
MeSH Terms: interventions — Cetylpyridinium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cetylpyridinium chloride/pH adjuster 1 (Active Comparator): A mouthwash contains cetylpyridinium chloride and pH adjuster 1.
  Interventions: Other: cetylpyridinium chloride
- Placebo 1 (Placebo Comparator): A mouthwash without cetylpyridinium chloride and pH adjuster 1
  Interventions: Other: cetylpyridinium chloride
- Cetylpyridinium chloride/pH adjuster 2 (Active Comparator): A mouthwash contains cetylpyridinium chloride and pH adjuster 2.
  Interventions: Other: cetylpyridinium chloride
- Placebo 2 (Placebo Comparator): A mouthwash without cetylpyridinium chloride and pH adjuster 2
  Interventions: Other: cetylpyridinium chloride

INTERVENTIONS:
Other: cetylpyridinium chloride — The mouthwash is used to see the effects on wound healing and the oral microbiome.

SUMMARY:
The purpose of this clinical research study is to investigate if mouthwashes to be tested can affect oral mucosal wound healing and change the oral microbiome (bacteria colonization) or expression of selected biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female volunteers 18-45 years of age.
2. Good general health.
3. Must sign informed consent form.
4. Minimum of 17 natural uncrowned teeth (excluding third molars) must be present.

Exclusion Criteria

1. Oral pathology, chronic disease, or history of allergy to testing product.
2. Medical condition which requires pre-medication prior to dental visits/procedures
3. Moderate or advanced periodontal disease (gum disease) or periodontal probing depths greater than 4 mm.
4. Five (5) or more decayed untreated dental sites at screening (cavities).
5. Impaired salivary function.
6. Use of medications that can currently affect salivary flow.
7. Use of anticonvulsants, antihistamines, antidepressants, sedatives, tranquilizers, antibiotics, antimicrobial, anti-inflammatory medication or daily analgesics within 30 days prior to the start of the study or scheduled to start such intake during the course of the study.
8. Ongoing use of medications known to affect the gingival tissues (i.e. calcium channel blockers, phenytoin, cyclosporine)
9. Pregnant or nursing women.
10. Participation in any other clinical study within 1 week prior to enrollment into this study.
11. Use of any tobacco products.
12. Subjects who must receive dental treatment during the study dates.
13. Presence of an orthodontic appliance that interferes with required clinical assessments.
14. History of allergy to common dentifrice ingredients.
15. Subjects who wear night guard, denture retainers
16. Not willing to abstain from eating crunchy (eg. Granola bars, popcorns, nuts etc) or spicy and hot foods/liquids during the study period;
17. Not willing to abstain from drinking citrus fluids, alcohol, and tea during the study period
18. Non English-speaking subjects

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Wound healing | 7 Days
  Images of the oral wounds will be taken before and after using the mouthwash treatment on days 1, 3, 5, and 7. The images will be taken on a digital camera. The wound sizes will be measured in mm2 using ImageJ software. The wound size will be measured at each time point and will be compared between a tested mouthwash and its placebo.
Microbiome | 5 Days
  Swabs will be collected from the hard palate on both the wounded and unwounded sides before and after injury and the mouthwash treatment at days 1, 3, 5, and 7. 16S rRNA sequencing will be performed to determine the bacteria microbiome. Correlations and relative abundance of bacteria will be compared at phylum and genus levels using bioinformatics tools between a mouthwash treated group and its placebo at different time points.

SECONDARY OUTCOMES:
Biomarker expression | 3 Days
  Real time polymerase chain reaction will be used to assess the mRNA expression of biomarkers in wound biopsy samples collected at days 1 and 3 post wounding and mouthwash treatment. The biomarkers include collagen I, collagen III, metalloproteinase-2, metalloproteinase-9, Interleukin-1β, Interleukin-6, and vascular endothelial growth factor. The fold changes of biomarker mRNA expression at each time point over the expression in unwounded tissues will be compared between a tested mouthwash and its placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Praveen Gajendrareddy, BDS, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- Clinical Research Center, College of Dentistry, University of Illinois Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No